CLINICAL TRIAL: NCT03244228
Title: A Two-part, Randomised, Double-blind, Placebo-controlled Single and Multiple Ascending Dose Study to Assess Safety, Pharmacokinetics and Pharmacodynamics of Oral HTL0016878 in Healthy Younger Adult and Elderly Subjects With a Randomised, Open-label, Crossover Arm to Assess the Effect of Food on Bioavailability of Oral HTL0016878.
Brief Title: A Two Part Study to Assess Safety, PK, PD, and Food Effect of Oral HTL0016878
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTL0016878-101; 2017-001385-26 (EudraCT Number); 16-028 (Other: HMR)
Record Dates: First submitted 2017-08-03; First posted 2017-08-09 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: First in human; Multiple ascending dose; Single ascending dose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1a SAD HTL0016878/Placebo (Experimental): In Part 1a, single ascending doses of HLT0016878 or matching placebo will be administered to groups of 12 subject each (9 active, 3 placebo). Each subject will have up to four treatment sessions separated by an appropriate wash-out. Healthy, young, male subjects.
  Interventions: Drug: HTL0016878; Drug: Placebo - Concentrate
- Part 1b single dose HTL0016878 (Experimental): In Part 1b, a single dose of HTL0016878 will be administered to 6 subjects on two occasions: once in the fasted and once the fed state. This will be open-label. Healthy, young, male or female subjects.
  Interventions: Drug: HTL0016878
- Part 1c single dose HTL0016878 (Experimental): In Part 1c, a single dose of HTL0016878 will be administered to up to 6 (optional up to 12) healthy elderly subjects This will be open-label. Healthy, elderly, male subjects.
  Interventions: Drug: HTL0016878
- Part 2a MAD HTL0016878/Placebo (Experimental): In Part 2a, multiple doses of HTL0016878 will be administered to up to 5 cohorts (N=8, 6 active, 2 placebo) during one study session of 7 days. Healthy, young, male or female subjects.
  Interventions: Drug: HTL0016878; Drug: Placebo - Concentrate
- Part 2b MAD HTL0016878/Placebo (Experimental): In Part 2b, multiple doses of HTL0016878 will be administered to up to 3 cohorts of healthy, elderly subjects (N=8, 6 active, 2 placebo) during one study session of 7 days. Healthy, young, male or female subjects.
  Interventions: Drug: HTL0016878; Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: HTL0016878 — Oral solution
Drug: Placebo - Concentrate — Matching placebo
  Arms: Part 1a SAD HTL0016878/Placebo; Part 2a MAD HTL0016878/Placebo; Part 2b MAD HTL0016878/Placebo

SUMMARY:
Phase 1, first in human, two-part, single centre, placebo-controlled, single and multiple ascending dose trial in healthy younger and elderly adult subjects, with an open-label, randomised, crossover arms to assess the effect of food on bioavailability.

DETAILED DESCRIPTION:
This is a first in human single and multiple ascending dose study with the objective to evaluate safety, tolerability, PK, PD, and food effect of HTL0016878 in healthy younger and elderly subjects. Part 1 will assess single doses of HTL0016878 and Part 2 will assess multiple doses of HTL0016878. Part 1 will be divided into 3 sub-parts: Part 1a will assess single ascending doses (SAD) of HTL0016878 in younger adult subjects, Part 1b will evaluate the effect of food on bioavailability of HTL0016878 and part 1c will investigate the effect of age on the PK of HTL0016878. Part 1c will only proceed after review of safety, tolerability and PK data from part 1a. Part 2 will be divided into 2 sub-parts to assess multiple ascending doses (MAD) of HTL0016878 in younger adult (part 2a) and elderly adult (part 2b) subjects. Part 2 will only proceed after review of safety, tolerability and PK data from Parts 1a, b and c.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive 18-55 year old (Parts 1a, 1b and 2a only) or 65+ year old (Parts 1c and 2b) male (all parts) or female (parts 1b, 2a and 2b only) volunteers with a body mass index 18-32kg/m².
* Healthy on the basis of a clinical history, physical examination, electrocardiogram (ECG), vital signs, heart rate (part 1a only), exercise history (part 1a only), and laboratory tests of blood and urine.
* Willingness to comply with requirements or the trial, including contraception requirements.
* Able to give fully informed consent.

Exclusion Criteria:

* Positive tests for hepatitis B & C, HIV
* severe adverse reaction to any drug
* sensitivity to trial medication
* drug or alcohol abuse
* smoking
* use of medication that inhibits CYP2D6 within previous 21 days or other prescribed and over-the-counter medication and herbal remedies within previous 21 days before dosing (with the exception of acetaminophen, contraceptive medications and hormone replacement therapy), unless the principal investigator (PI) considers that it would not interfere with trial
* participation in other clinical trials of unlicensed medicines in the previous 3 months, or regularly take part in more than 4 studies a year
* loss of more than 500 mL blood in the previous 3 months
* vital signs, QTcF interval or laboratory values outside the acceptable range
* poor metabolizers of CYP2D6 (apart from one optional cohort in Part 1a, which may enrol poor metabolizers only)
* clinically relevant abnormal findings at the screening assessment
* acute or chronic illness
* history of epilepsy or seizures
* clinically relevant abnormal medical history or concurrent medical condition
* disease associated with cognitive impairment and/or psychosis
* recent history of suicidal thoughts or ideation, or insomnia
* excessive use of caffeine containing beverages, exceeding 8 cups of coffee or equivalent/day and the inability to refrain from the use of caffeine containing beverages whilst on the ward
* consumption of cranberry, pomegranate, star fruit, grapefruit, pomelos, exotic citrus fruits or Seville oranges (including marmalade and juices made from these fruits) within 3 days before admission; possibility that volunteer will not cooperate
* pre-menopausal females who are pregnant or lactating, or who are sexually active and not using a reliable method of contraception
* Objection by the GP.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) | Baseline up to 14 days post dose
  Safety and Tolerability
Physical examinations | Baseline up to 14 days post dose
  Safety and Tolerability
vital signs (Heart Rate and Blood pressure) | Baseline up to 14 days post dose
  Safety and Tolerability
Laboratory safety assessment | Baseline up to 14 days post dose
  Safety and Tolerability
ECG | Baseline up to 14 days post dose
  Safety and Tolerability
Columbia- suicide severity rating scale (C-SSRS) | Baseline up to 14 days post dose
  Safety and Tolerability

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of HTL0016878 | Baseline up to 14 days post dose
  Pharmacokinetics
Time to Maximum plasma concentration (Tmax) of HTL0016878 | Baseline up to 14 days post dose
  Pharmacokinetics
Area under the curve of HTL0016878 | Baseline up to 14 days post dose
  Pharmacokinetics
Half-life (t1/2) of HTL0016878 | Baseline up to 14 days post dose
  Pharmacokinetics
Amount excreted in urine (Ae) of HTL0016878 | Baseline up to 14 days post dose
  Pharmacokinetics
Fraction of dose eliminated unchanged on urine (fe/F) of HTL0016878 | Baseline up to 14 days post dose
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, Hammersmith, United Kingdom

IPD SHARING:
Plan to Share IPD: No